CLINICAL TRIAL: NCT05030129
Title: An Exploratory Single Blind Study of Ergoloid Mesylates, 5-Hydroxytryptophan, and the Combination in Adult Males With Fragile X Syndrome
Brief Title: ERG/5-HTP in Fragile X Syndrome (FXS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Berry-Kravis (Other)
Collaborators: FRAXA Research Foundation (Other); Purposeful IKE (Industry)
Responsible Party: Sponsor-Investigator, Elizabeth Berry-Kravis, Professor, Department of Pediatrics, Neurological Sciences, Biochemistry, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ORA 21051102
Record Dates: First submitted 2021-08-05; First posted 2021-09-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — 5-Hydroxytryptophan; Ergoloid Mesylates

STUDY DESIGN:
Intervention Model Description: This study will use a single-blind, 4-period sequential design. Fifteen participants with Fragile X Syndrome ages 18-45 years will enter a Screening period of up to 28 days followed by four 4 week single-blind treatment periods (summarized below).
  * Period 1: Ergoloid mesylates 1 mg and matching placebo for 5-Hydroxytryptophan 100 mg, taken three times per day
  * Period 2: Ergoloid mesylates 1 mg and 5-Hydroxytryptophan 100 mg, taken three times per day
  * Period 3: 5-Hydroxytryptophan 100 mg and matching placebo for Ergoloid mesylates 1mg, taken three times per day
  * Period 4: Matching placebo for Ergoloid mesylates 1mg and matching placebo for 5- Hydroxytryptophan 100mg, taken three times per day
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a single-blind study, meaning the participant and his family/caregivers will not know what drug or combination the participant is receiving during each time period. The investigator and study coordinator will know what drug the participant is taking. The remainder of the study team performing assessments such as the Vineland, eye tracking, ERP, Toolbox, and the KiTAP will not know the type of treatment the patient is on when testing is done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ergoloid mesylates (EM) (Experimental): During treatment period 1, subjects will receive EM 1 mg (Medisca) and matching placebo for 5-HTP 100mg (ascorbic acid powder). One of each capsule (both size 00) will be taken three times per day for four weeks.
  Interventions: Drug: Ergoloid Mesylates; Drug: Matching placebo for 5-Hydroxytryptophan
- Ergoloid mesylates (EM) and 5-hydroxytryptophan (5-HTP) (Experimental): During treatment period 2, subjects will receive EM 1 mg (Medisca) and 5-HTP 100 mg (5-HTP, Basic Vitamins). One of each capsule (both size 00) will be taken three times per day for four weeks.
  Interventions: Drug: 5-Hydroxytryptophan; Drug: Ergoloid Mesylates
- 5-hydroxytryptophan (5-HTP) (Experimental): During treatment period 3, subjects will receive 5-HTP 100 mg (5-HTP, Basic Vitamins) and matching placebo for EM 1 mg (ascorbic acid powder). One of each capsule (both size 00) will be taken three times per day for four weeks.
  Interventions: Drug: 5-Hydroxytryptophan; Drug: Matching placebo for Ergoloid mesylates
- Placebo (Placebo Comparator): During treatment period 4, subjects will receive matching placebo for EM 1mg (ascorbic acid powder) and matching placebo for 5-Hydroxytryptophan 100mg (ascorbic acid powder). One of each capsule (both size 00) will be taken three times per day for four weeks.
  Interventions: Drug: Matching placebo for Ergoloid mesylates; Drug: Matching placebo for 5-Hydroxytryptophan

INTERVENTIONS:
Drug: 5-Hydroxytryptophan — 5-HTP will be over-encapsulated in identical size 00 capsules. During the 5-HTP Treatment Period (Period 3) and 5-HTP/EM Treatment Period (Period 2), subjects will take 1 capsule of 5-HTP 3 times per day.
  Other Names: 5-HTP, Basic Vitamins
  Arms: 5-hydroxytryptophan (5-HTP); Ergoloid mesylates (EM) and 5-hydroxytryptophan (5-HTP)
Drug: Ergoloid Mesylates — Ergoloid mesylates 1 mg will be mixed with methyl cellulose and placed in a size 00 capsule. During the EM Treatment Period (Period 1) and 5-HTP/EM Treatment Period (Period 2), subjects will take 1 capsule of EM 3 times per day.
  Other Names: Medisca
  Arms: Ergoloid mesylates (EM); Ergoloid mesylates (EM) and 5-hydroxytryptophan (5-HTP)
Drug: Matching placebo for Ergoloid mesylates — Matching placebo for Ergoloid mesylates will be ascorbic acid powder in identical size 00 capsules. During the 5-HTP Treatment Period (Period 3) and Placebo Treatment Period (Period 4), subjects will take 1 capsule of matching placebo for EM 3 times per day.
  Arms: 5-hydroxytryptophan (5-HTP); Placebo
Drug: Matching placebo for 5-Hydroxytryptophan — Matching placebo for 5-Hydroxytryptophan will be ascorbic acid powder in identical size 00 capsules. During the EM Treatment Period (Period 2) and Placebo Treatment Period (Period 4), subjects will take 1 capsule of matching placebo for 5-HTP 3 times per day.
  Arms: Ergoloid mesylates (EM); Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and efficacy of Ergoloid mesylates (EM) and 5-hydroxytryptophan (5-HTP) and the combination (EM + 5-HTP) compared to placebo in males aged 18-45 years old with Fragile X Syndrome.

DETAILED DESCRIPTION:
This single-center, Phase 2, single-blind, 4-period sequential study will enroll 15 males Fragile X Syndrome, ages 18-45 years old.

The study will begin with a Screening period of up to 28 days. During screening, participants and their parent/legal authorized guardian, if indicated, will review and sign an Informed Consent/Assent form prior to any study procedures being performed. Following confirmation of a prior diagnosis for Fragile X, information will be collected to further assess their eligibility.

Participants who meet entry criteria and agree to participate will proceed to a Baseline visit. At the Baseline visit (Period 1/Day 1), cognitive, behavioral, ERP and eye tracking assessments will be performed to assess current functioning.

The Baseline visit will be followed by four 4-week single-blind treatment periods. During treatment periods, participants will be placed on a different treatment regimen every 4 weeks (listed below). Throughout all 4 periods, participants will take two identical capsules three times a day. If only taking one study drug, they will take one placebo pill with the drug at each dose, and in period 4, they will take two placebo pills at each dose.

* Period 1: Ergoloid mesylates (EM) 1 mg three times per day for 4 weeks
* Period 2: Ergoloid mesylates (EM) 1 mg TID and 5-hydroxytryptophan (5-HTP) 100 mg three times per day for 4 weeks
* Period 3: 5-hydroxytryptophan (5-HTP) 100 mg three times per day for 4 weeks
* Period 4: Placebo three times per day for 4 weeks

Participants will return to the clinic at the end of each treatment period at weeks 4, 8, 12, and 16 and cognitive and behavioral evaluations will be repeated at these clinic visits. Safety and tolerability assessments will include adverse event monitoring, vital signs, blood chemistry and hematology, and urinalysis. Additionally, participants will be monitored for adverse events via a telephone call at the end of Week 1 of each Period, and one week following completion of Period 4 or following early discontinuation. Total study participation will last up to 21 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18 to 45 years, inclusive.
2. Participant has Fragile X Syndrome with a molecular genetic confirmation of the full Fragile X Mental Retardation (FMR1) mutation (≥200 CGG repeats).
3. Current treatment with no more than 3 prescribed psychotropic medications. Anti-epileptic medications are permitted and are not counted as psychotropic medications if they are used for treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications.
4. Permitted concomitant psychotropic medications must be at a stable dose and dosing regimen for at least 2 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
5. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
6. Participants with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure-free for 3 months preceding screening, or must be seizure-free for 3 years if not currently receiving anti-epileptics.
7. Behavioral and therapy treatments/interventions must be stable for 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication, and throughout the study. Minor changes in hours or times of therapy that are not considered clinically significant will not be exclusionary. Changes in therapies provided through a school program, due to school vacations, are allowed.
8. Participant must be willing to practice barrier methods of contraception while on study, if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.
9. Participant has a parent, legal authorized guardian or consistent caregiver.
10. Participant and caregiver are able to attend the clinic regularly and reliably.
11. Participant is able to swallow capsules.
12. For participants who are not their own legal guardian, participant's parent/legal authorized guardian is able to understand and sign an informed consent form to participate in the study.
13. If participant is his own legal guardian, he can understand and sign informed consent to participate in the study.
14. If participant is not their own legal guardian, the participant provides assent for participation in the study, if the participant has the cognitive ability to provide assent.

Exclusion Criteria:

1. History of, or current cardiovascular, renal, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cerebrovascular, or other systemic disease that would place the participant at risk or potentially interfere with the interpretation of the safety, tolerability, or efficacy of the study medication.

   Common diseases such as mild hypertension, well-controlled type 2 diabetes mellitus (hemoglobin A1C [Hgb A1C] <6.5%), etc. are allowed per the investigator's judgment as long as they are stable and controlled by medical therapy that is constant for at least 4 weeks before randomization.
2. Clinically significant abnormalities, in the investigator's judgment, in safety laboratory tests, vital signs, as measured during Screening.
3. History of substance abuse within the past year, according to investigator assessment.
4. Use of CYP3A4 inhibitors, beta-blockers, MAO inhibitors or triptans at any time during participation in the study.
5. Significant hearing or visual impairment that may affect the participant's ability to complete the test procedures.
6. Concurrent major psychiatric condition (e.g., Major Depressive Disorder, Schizophrenia or Bipolar Disorder) as diagnosed by the investigator. Participants with additional diagnosis of Autism Spectrum Disorder or Anxiety Disorder will be allowed as these are characteristics of FXS.
7. Participant has active diseases that would interfere with participation, such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
8. Participant is planning to commence psychotherapy or cognitive behavior therapy (CBT) during the period of the study or had begun psychotherapy or CBT within 4 weeks prior to Screening.
9. Participant has participated in another clinical trial within the 30 days preceding Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Males With Fragile X Syndrome: Fifteen participants with Fragile X syndrome ages 18-45 years old will be enrolled in this single-blind study. Eligible participants will be started on EM for 4 weeks in Treatment Period 1, then will take EM and 5-HTP for 4 weeks in Treatment Period 2, then, 5-HTP for 4 weeks in Treatment Period 3, then placebo for 4 weeks in Treatment Period 4.
Period: Screening Period
Arm/Group | Adult Males With Fragile X Syndrome
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 1: EM & Placebo
Arm/Group | Adult Males With Fragile X Syndrome
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 2: EM & 5-HTP
Arm/Group | Adult Males With Fragile X Syndrome
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 3: 5-HTP & Placebo
Arm/Group | Adult Males With Fragile X Syndrome
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 4: Placebo
Arm/Group | Adult Males With Fragile X Syndrome
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Males With Fragile X Syndrome
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
KiTAP Executive Battery - Alertness Subscore (Reaction Time) [Mean (Full Range); unit: milliseconds] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The alertness subtest requires subjects to tap a button every time a stimulus appears on the screen. Mean reaction time was measured over 90 seconds. A lower reaction time indicates better performance.
  milliseconds | 482.7857143 [112 to 1297]
KiTAP Executive Battery Distractibility Subtest - Total Number of Correct Responses [Mean (Full Range); unit: Correct Responses] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The distractibility subtest measures how easily the subject is distracted by extraneous stimuli. This subtest requires subjects to tap a button when a target stimulus appears on the screen while ignoring distracters that appear shortly before the stimulus. A high mean number of correct responses and low mean number of errors over the 3 minutes indicates better performance.
  Correct Responses | 11.78 [1 to 18]
KiTAP Executive Battery Distractibility Subtest - Total Number of Errors [Mean (Full Range); unit: Errors] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The distractibility subtest measures how easily the subject is distracted by extraneous stimuli. This subtest requires subjects to tap a button when a target stimulus appears on the screen while ignoring distracters that appear shortly before the stimulus. A high mean number of correct responses and low mean number of errors over the 3 minutes indicates better performance.
  Errors | 6.214285714 [0 to 19]
KiTAP Executive Battery Flexibility Subtest - Total Number of Correct Responses [Mean (Full Range); unit: Correct Responses] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The flexibility subtest measures the subject's ability to be flexible about shifting from one response type to another. This subtest is 2 minutes long and requires subjects to alternate between identifying blue and green dragons which seem on random sides of the screen by tapping one of two buttons. A high mean number of correct responses and low mean number of errors indicates better performance.
  Correct Responses | 14.64 [8 to 26]
KiTAP Executive Battery Flexibility Subtest - Total Number of Errors [Mean (Full Range); unit: Errors] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The flexibility subtest measures the subject's ability to be flexible about shifting from one response type to another. This subtest is 2 minutes long and requires subjects to alternate between identifying blue and green dragons which seem on random sides of the screen by tapping one of two buttons. A high mean number of correct responses and low mean number of errors indicates better performance.
  Errors | 12.29 [6 to 18]
KiTAP Test of Attentional Performance Go-NoGo Subtest - Total Number of Correct Responses [Mean (Full Range); unit: Correct Responses] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The Go-NoGo subtest measures a subject's impulsivity by requiring subjects to tap a button when the target stimulus is presented, while refraining from hitting the button for the non-target stimulus. This subtest takes place over 2 minutes 30 seconds. A high mean number of correct responses and a low mean number of errors indicates better performance.
  Correct Responses | 14.86 [3 to 20]
KiTAP Test of Attentional Performance Go-NoGo Subtest - Total Number of Errors [Mean (Full Range); unit: Errors] — The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The Go-NoGo subtest measures a subject's impulsivity by requiring subjects to tap a button when the target stimulus is presented, while refraining from hitting the button for the non-target stimulus. This subtest takes place over 2 minutes 30 seconds. A high mean number of correct responses and a low mean number of errors indicates better performance.
  Errors | 9.57 [0 to 21]
Clinical Global Impression - Severity (CGI-S) Scale Overall Score [Count of Participants; unit: Participants] — The Clinical Global Impression-Severity (CGI-S) is a global measure to provide a clinical judgment of a participant's overall condition based on a trained clinician's assessment of cognition, behavior and activities of daily living. The clinician compares the subject with individuals of the same age and sex. The assessment of severity is with a 7-point scale: 1, not ill; 2, very mild; 3, mild; 4, moderate; 5, marked; 6, severe; 7, extremely severe.
  Participants
    Extremely Severe | 0
    Severe | 0
    Marked | 5
    Moderate | 8
    Mild | 2
    Very Mild | 0
    Not Ill | 0
Aberrant Behavior Checklist (ABC) Subscores [Mean (Full Range); unit: scores on a scale] — This assessment is a parent/caregiver-rated scale with six subscales to assess irritability, stereotypes, lethargy, hyperactivity, inappropriate speech, and social avoidance, using ABC-FX factoring system. The range of possible scores are irritability (0-54), lethargy (0-39), stereotypes (0-18), hyperactivity (0-30), inappropriate speech (0-12), and social avoidance (0-12). Mean score for each subscale was calculated. Lower scores on each subscale indicate fewer aberrant behaviors (better functioning).
  scores on a scale
    Irritability Subscale | 6.666666667 [0 to 24]
    Lethargy Subscale | 4.8 [0 to 25]
    Stereotypes Subscale | 2.666666667 [0 to 12]
    Hyperactivity Subscale | 4.733333333 [0 to 12]
    Inappropriate Speech Subscale | 4.4 [2 to 12]
    Social Avoidance Subscale | 4.133333333 [0 to 12]
Anxiety, Depression, and Mood Scale (ADAMS) Subscores [Mean (Full Range); unit: scores on a scale] — The ADAMS is a parent/caregiver rated scale with five sub-scores to assess manic/hyperactive behavior, depressed mood, social avoidance, general anxiety, and obsessive/compulsive behavior. The range of possible scores for each subscale is 0-21. Lower mean scores on each subscale indicate better functioning.
  scores on a scale
    Manic/Hyperactive Behavior Subscore | 5.333333333 [1 to 11]
    Depressed Mood Subscore | 3.2 [0 to 12]
    Social Avoidance Subscore | 8 [1 to 21]
    General Anxiety Subscore | 6.666666667 [2 to 13]
    Obsessive/Compulsive Behavior Subscore | 1.866666667 [0 to 6]
Vineland-3 Adaptive Behavior Scale (VABS-3) - Subdomain Growth Scale Values [Mean (Full Range); unit: score on a scale] — VABS-3 is a clinician-administered standardized interview. For this study, we collected data in domains of communication (receptive & written language), daily living skills (domestic & community skills), & socialization (interpersonal relationships, play & leisure time, & coping abilities). Mean growth scale value (GSV) for each subdomain is reported. The possible GSVs for each subdomain are receptive (10-162), written (10-163), domestic (10-110), community (10-136), interpersonal (10-152), play and leisure (10-164), & coping skills (10-120). Higher GSVs indicate better functioning.
  score on a scale
    Receptive Communication Subdomain | 126.5 [95 to 151]
    Written Communication Subdomain | 91 [47 to 115]
    Daily Living Skills - Community Subdomain | 67.35714286 [46 to 82]
    Daily Living Skills - Domestic Subdomain | 60.92857143 [44 to 81]
    Social - Interpersonal Relationships Subdomain | 101.7857143 [79 to 129]
    Social - Play and Leisure Subdomain | 105.9230769 [83 to 120]
    Social - Coping Skills Subdomain | 69.5 [53 to 82]
NIH Toolbox Cognitive Battery for Intellectual Disabilities (NIH-TCB) Total Cognition Score [Mean (Full Range); unit: score on a scale] — The NIH-TCB is a battery of extensively validated computer-administered cognitive tests. The battery produces fluid and crystallized composite scores. The Total Cognition Composite Score is found by converting raw fluid and crystallized cognition scores to standard scores, averaging the these two scaled scores, then deriving standard scores based on this new distribution. Scores range from 0-140. The normative mean of the uncorrected score is 100 and the standard deviation is 15. A higher mean total cognition uncorrected composite score indicates better performance.
  score on a scale | 57.3 [35 to 78]
Visual Analog Scale (VAS) Assessment Domain Scores [Mean (Full Range); unit: score on a scale] — In an attempt to measure the level of behavioral difficulty experienced by the parent/caregiver with respect to the child with FXS, the VAS allows parents to mark on a visual line measuring 10 cm with one side marked "worst behavior" and the other side marked "best behavior." The caregiver rates the participant's behavior with respect to three domains: daily functioning, anxiety/irritability and language. Distances closer to 10 cm are considered worse behavior and distances closer to 0 cm are considered better behavior.
  score on a scale
    Target Language Issues | 5.241333333 [0 to 9.6]
    Daily Function Issues | 6.11 [1.91 to 9.7]
    Anxiety or Irritability Issues | 5.426666667 [0.5 to 9.9]
Event-Related Potentials (ERP) - Gamma Band Absolute Power at Resting State (Frontal) [Mean (Standard Deviation); unit: V^2/Hz] — Event-Related Potentials (ERPs) enable extraction of neural responses associated with specific sensory, cognitive, or motor events from an overall EEG. Gamma 1 and gamma 2 waves were measured for various parts of the brain at a resting state. FXS patients have typically been found to exhibit greater gamma frequency band power than typically developing controls, which may be related to social and sensory processing difficulties. Therefore, lower gamma band power would indicate better functioning.
  V^2/Hz
    Gamma 1 (30-55 Hz) Absolute Power | 0.047656355 (0.018258564)
    Gamma 2 (65-80 Hz) Absolute Power | 0.026220458 (0.011025469)
Event-Related Potential (ERP) Components in Response to Standard Tones [Mean (Standard Deviation); unit: μV*seconds] — Event-Related Potentials (ERPs) enable extraction of neural responses associated with specific sensory, cognitive, or motor events from an overall EEG. Auditory stimuli are presented and EEG events are assessed in relation to timing of the stimuli. The area under the curve was measured for different components of the ERP including P1 and P2 (positive components) and N1 and N2 (negative components) and the average area was reported.
  μV*seconds
    P1 Component | 0.01171 (0.010617538)
    P2 Component | 0.0345626 (0.032675507)
    N1 Component | 0.0164247 (0.022616337)
    N2 Component | 0.0360871 (0.041661709)
Event-Related Potentials - Frontal Alpha Asymmetry at Resting State [Mean (Standard Deviation); unit: unitless] — ERP data was collected while the subject was in a resting state. Frontal alpha asymmetry measures differences in alpha activity level of the right and left hemisphere of the frontal lobe of the brain. Higher alpha asymmetry scores indicate greater alpha power in the right hemisphere, which corresponds to increased neural activity in the left hemisphere. High activity of the left frontal lobe is hypothesized to correspond with approach behaviors, and high activity of the right frontal lobe is thought to correspond to withdrawal behaviors.
  unitless | -0.049005225 (0.326769814)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability - Number of Treatment-Emergent Adverse Events
Description: Adverse Events (AEs), including clinically meaningful laboratory abnormalities and significant behavioral changes will be recorded from the time of the subject's first dose of study drug to the end of the study (Week 17) or longer if needed. Adverse events will be assessed at each visit as well as during each phone call and will be tabulated for each treatment period.
Time Frame: Baseline through Week 17
Population: The Safety population will include all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Adverse Events
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Number of Adverse Events | 2 | 1 | 1 | 3

2. Primary Outcome: Safety and Tolerability - Severity of Treatment Emergent Adverse Events
Description: Adverse Events (AEs), including clinically meaningful laboratory abnormalities and significant behavioral changes will be tabulated for each treatment period.
  The Investigator is responsible for assessing the severity (intensity) of each adverse event as mild, moderate, or severe according to the following definitions:
  Mild - An event that is easily tolerated and generally not interfering with normal daily activities. Moderate - An event that is sufficiently discomforting to interfere with normal daily activities. Severe - An event that is incapacitating with inability to work or perform normal daily activities.
Time Frame: Baseline through Week 17
Population: The Safety population will include all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Adverse Events
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Number of Adverse Events
  Mild | 2 | 1 | 1 | 2
  Moderate | 0 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in KiTAP Executive Battery - Alertness Subscore (Reaction Time)
Description: The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The alertness subtest requires subjects to tap a button every time a stimulus appears on the screen. KiTAP was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). Mean reaction time was measured over 90 seconds and change from baseline was calculated. A lower reaction time (net decrease in reaction time) indicates better performance.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: Intent to treat (ITT) efficacy population, which will include all participants who received at least one dose of treatment and returned for at least one follow-up visit.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
milliseconds | -78.2678 (107.4594) | -0.52675 (107.4594) | 14.3989 (109.7533) | 31.48097 (109.7533)

4. Secondary Outcome: Change From Baseline in Total Number of Correct Responses on KiTAP Executive Battery Distractibility Subtest
Description: The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The distractibility subtest measures how easily the subject is distracted by extraneous stimuli. This subtest requires subjects to tap a button when a target stimulus appears on the screen while ignoring distracters that appear shortly before the stimulus. KiTAP was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). Mean number of correct responses and errors were recorded, and change from baseline was calculated. For the distractability subtest, a higher mean number of correct responses and lower mean number of errors over the 3 minutes indicates better performance.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: Intent to treat (ITT) efficacy population, which includes all participants who received at least one dose of treatment and returned for at least one follow-up visit.
Measure: Mean (Standard Error); unit: Correct Responses
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Correct Responses | 2.142857 (2.9003) | -3.1705358 (2.9201) | 0.8607271 (2.9201) | -4.0571867 (2.9201)

5. Secondary Outcome: Change From Baseline in Total Number of Errors on KiTAP Executive Battery Distractibility Subtest
Description: as for outcome 4
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Errors
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Errors | 2.64285 (2.7233) | 0.53599 (2.8155) | 0.79141 (2.8155) | -1.9874 (2.7474)

6. Secondary Outcome: Change From Baseline in Total Number of Correct Responses on KiTAP Executive Battery Flexibility Subtest
Description: The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The flexibility subtest measures the subject's ability to be flexible about shifting from one response type to another. This subtest is 2 minutes long and requires subjects to alternate between identifying blue and green dragons which seem on random sides of the screen by tapping one of two buttons. KiTAP was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). Mean number of correct responses and errors were recorded and change from baseline was calculated. For the flexibility subtest, a higher mean number of correct responses and lower mean number of errors indicates better performance.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Correct Responses
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Correct Responses | -1.928571 (1.1029) | -1.452112 (1.1124) | -3.340254 (1.1124) | -1.237821 (1.1124)

7. Secondary Outcome: Change From Baseline in Total Number of Errors on KiTAP Executive Battery Flexibility Subtest
Description: as for outcome 6
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Errors
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Errors | 1.5 (0.7120) | 1.93979 (0.7178) | 2.05569 (0.7178) | 1.56290 (0.7178)

8. Secondary Outcome: Change From Baseline in Total Number of Correct Responses on KiTAP Test of Attentional Performance Go-NoGo Subtest
Description: The KiTAP is a computerized executive function battery that consists of eight nonverbal subtests measuring different basal as well as higher-order components of attention and executive functioning. The Go-NoGo subtest measures a subject's impulsivity by requiring subjects to tap a button when the target stimulus is presented, while refraining from hitting the button for the non-target stimulus. KiTAP was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). This subtest takes place over 2 minutes 30 seconds. Mean number of correct responses and errors were recorded, and change from baseline was calculated. For the Go-NoGo subtest, a higher mean number of correct responses and a lower mean number of errors indicates better performance.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: The primary efficacy population will be the intent to treat (ITT) efficacy population, which will include all participants who received at least one dose of treatment and returned for at least one follow-up visit.
Measure: Mean (Standard Error); unit: Correct Responses
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Correct Responses | 0.3966214 (1.5644) | 1.8198629 (1.5962) | 0.4632881 (1.5644) | -1.1383753 (1.5962)

9. Secondary Outcome: Change From Baseline in Total Number of Errors on KiTAP Test of Attentional Performance Go-NoGo Subtest
Description: as for outcome 8
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Errors
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Errors | -0.1177 (1.5019) | 0.55828 (1.5335) | 0.28221 (1.5019) | 0.73542 (1.5335)

10. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity Scale Overall Score
Description: The Clinical Global Impression-Severity (CGI-S) is a global measure to provide a clinical judgment of a participant's overall condition based on a trained clinician's assessment of cognition, behavior and activities of daily living. The clinician compares the subject with individuals of the same age and sex. The assessment of severity is with a 7-point scale: 1, not ill; 2, very mild; 3, mild; 4, moderate; 5, marked; 6, severe; 7, extremely severe. A net decrease in severity score over time indicates a positive outcome.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
scores on a scale | -0.06667 (0.0805) | -0.06667 (0.0805) | -0.06667 (0.0805) | -0.06667 (0.0805)

11. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Subscores
Description: This assessment is a parent/caregiver-rated scale with six subscales to assess irritability, stereotypes, lethargy, hyperactivity, inappropriate speech, and social avoidance, using ABC-FX factoring system. The ABC was was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). Mean score for each subscale was measured and change from baseline was calculated. Lower mean scores on each subscale indicate fewer aberrant behaviors (better functioning).The range of possible scores on each subscale are irritability (0-54), lethargy (0-39), stereotypes (0-18), hyperactivity (0-30), inappropriate speech (0-12), and social avoidance (0-12).
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  Irritability Subscale | -2.59088 (0.9919) | -2.36774 (0.9919) | -2.53333 (0.9706) | -2.13333 (0.9706)
  Lethargy Subscale | -0.86667 (0.8081) | -0.34695 (0.8258) | -0.79147 (0.8258) | -1.8 (0.8081)
  Stereotypes Subscale | -0.73333 (0.5678) | -0.82132 (0.5801) | -1.06667 (0.5678) | -0.8 (0.5678)
  Hyperactivity Subscale | -0.6 (0.5241) | -1.31738 (0.5355) | -1.46667 (0.5241) | -1.4 (0.5241)
  Inappropriate Speech Subscale | -0.53333 (0.3355) | -0.9934 (0.3429) | -1.46667 (0.3355) | -1.46667 (0.3355)
  Social Avoidance Subscale | -0.73333 (0.3362) | -0.64283 (0.3520) | -0.50848 (0.3436) | -0.4 (0.3362)

12. Secondary Outcome: Change From Baseline in Anxiety, Depression, and Mood Scale (ADAMS) Subscores
Description: The ADAMS is a parent/caregiver rated scale with five subscores to assess manic/hyperactive behavior, depressed mood, social avoidance, general anxiety, and obsessive/compulsive behavior. The ADAMs was completed at Baseline as well as Week 4, Week 8, Week 12, and Week 16 (the end of each treatment period). Mean score for each subscale was recorded, and change from baseline was calculated for each subscore. The range of possible scores for each subscale is 0-21. Lower mean scores on each subscale indicate better functioning.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  Manic/Hyperactive Behavior Total Score | -1.4 (0.4076) | -1.7333 (0.4076) | -2.26667 (0.4076) | -1.8 (0.4076)
  Depressed Mood Total Score | -1.13333 (0.6433) | -0.06667 (0.6433) | -1.13333333 (0.6433) | -1.6 (0.6433)
  Social Avoidance Total Score | -1.733333 (0.6911) | -1.333333 (0.6911) | -2.666667 (0.6911) | -1.866667 (0.6911)
  General Anxiety Total Score | -1.533333 (0.6770) | -1.8 (0.6770) | -2.946642 (0.6770) | -2.266667 (0.6770)
  Obsessive/Compulsive Behavior Total Score | -0.13333333 (0.3792) | 0.06666667 (0.3792) | -0.2 (0.3792) | -0.4 (0.3792)

13. Secondary Outcome: Change From Baseline on Vineland-3 Adaptive Behavior Scale - Subdomain Growth Scale Values
Description: VABS-3 is a clinician-administered standardized interview. For this study, we collected data in domains of communication (receptive & written language), daily living skills (domestic & community skills), & socialization (interpersonal relationships, play & leisure time, & coping abilities). This assessment was administered at Baseline as well as at Week 4, Week 8, Week 12, and Week 16 (end of each treatment period). Mean growth scale value (GSV) for each subdomain was recorded at each time point and change from baseline was calculated. The possible GSVs for each subdomain are receptive (10-162), written (10-163), domestic (10-110), community (10-136), interpersonal (10-152), play and leisure (10-164), & coping skills (10-120). Higher GSVs for each subdomain indicate better functioning.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  Receptive Communication Subdomain | 0.3603766 (3.0827) | 4.4457568 (2.9079) | 3.9678919 (2.6167) | 5.2990546 (2.7389)
  Written Communication Subdomain | 3.926537 (2.6030) | 3.915339 (2.4556) | 5.287075 (2.2088) | 5.051526 (2.3123)
  Daily Living Skills - Community Subdomain | 2.2145 (1.9946) | 3.437951 (1.8816) | 2.733986 (1.6921) | 4.313574 (1.7715)
  Daily Living Skills - Domestic Subdomain | -1.940166 (2.4600) | 1.421966 (2.3207) | 5.013375 (2.0873) | 5.501518 (2.1852)
  Social - Interpersonal Relationships Subdomain | 6.01876 (2.3460) | 6.042022 (2.2132) | 6.664025 (1.9898) | 5.801988 (2.0834)
  Social - Play and Leisure Subdomain | -10.989137 (6.4126) | -3.47187 (6.0588) | -1.203629 (5.5469) | 5.592143 (5.8006)
  Social - Coping Skills Subdomain | 1.460214 (2.8857) | 2.756048 (2.7214) | 2.077872 (2.4548) | 7.090882 (2.5673)

14. Secondary Outcome: Change From Baseline in NIH Toolbox Cognitive Battery for Intellectual Disabilities (NIH-TCB) Total Cognition Score
Description: The NIH-TCB is a battery of extensively validated computer-administered cognitive tests. The NIH-TCB includes 7 evaluations measuring cognitive flexibility, inhibition & visual attention, episodic memory, immediate recall & sequencing of different visually & orally presented stimuli, processing speed, recognition of letters and words, & receptive vocabulary. This assessment was administered at Baseline as well as at Week 4, Week 8, Week 12, and Week 16 (end of each treatment period). This battery produces fluid and crystallized cognition composite scores. The Total Cognition Composite Score is found by converting raw fluid and crystallized scores to standard scores, averaging these two scores, then deriving standard scores based on this new distribution. Scores range from 0-140. The normative mean of the uncorrected standard score is 100 and the standard deviation is 15. A higher mean total cognition composite score indicates better performance.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 4
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
scores on a scale | 2.10074 (4.5470) | -9.156292 (6.9968) | -4.734578 (5.0309) | -2.531407 (4.1965)

15. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Assessment Domain Scores
Description: IIn an attempt to measure the level of behavioral difficulty experienced by the parent/caregiver with respect to the child with FXS, the VAS allows parents to mark on a visual line measuring 10 cm with one side marked "worst behavior" and the other side marked "best behavior." The caregiver rated the participant's behavior with respect to three domains: daily functioning, anxiety/irritability and language. Distances closer to 10 cm are considered worse behavior and distances closer to 0 cm are considered better behavior. Average distance of the mark was recorded for each domain at Baseline then again at Week 4, Week 8, Week 12, and Week 16 (end of each treatment period). Change from baseline was calculated for each domain. Lower scores indicate a better outcome (closer distance to best behavior side).
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  Target Language Issues | 0.9786667 (0.5869) | 0.9786667 (0.5869) | 0.712 (0.5869) | 0.5253333 (0.5869)
  Daily Function Issues | 0.6833333 (0.5763) | 0.8433333 (0.5763) | 0.6566667 (0.5763) | 0.93 (0.5763)
  Anxiety or Irritability Issues | 0.2533333 (0.6165) | 1.1233333 (0.6165) | 0.6433333 (0.6165) | -0.2933333 (0.6165)

16. Secondary Outcome: Event-Related Potentials (ERP) - Gamma Band Absolute Power at Resting State (Frontal)
Description: Event-Related Potentials (ERPs) enable extraction of neural responses associated with specific sensory, cognitive, or motor events from an overall EEG. Gamma 1 and gamma 2 waves were measured for various parts of the brain at a resting state. ERP was performed at Baseline as well as at Week 4, Week 8, Week 12, Week 16 (at the end of each treatment period). Mean power of gamma 1 and gamma 2 bands, measured by frontal EEG leads, was recorded for each time point and change from baseline was calculated. FXS patients have typically been found to exhibit greater gamma frequency band power than typically developing controls, which may be related to social and sensory processing difficulties. Therefore, lower gamma band power would indicate better functioning.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: V^2/Hz
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
V^2/Hz
  Gamma 1 (30-55 Hz) Absolute Power | 0.054717778 (0.009638014) | 0.051050595 (0.006690128) | 0.061321956 (0.007923461) | 0.050649034 (0.010533546)
  Gamma 2 (65-80 Hz) Absolute Power | 0.027005807 (0.005267368) | 0.025525849 (0.004251649) | 0.031589661 (0.004834075) | 0.025235128 (0.004757463)

17. Secondary Outcome: Event-Related Potentials (ERP) Components in Response to Standard Tones
Description: Event-Related Potentials (ERPs) enable extraction of neural responses associated with specific sensory, cognitive, or motor events from an overall EEG. Auditory stimuli are presented and EEG events are assessed in relation to timing of the stimuli. ERP was performed at Baseline as well as at week Week 4, Week 8, Week 12, Week 16 (end of each treatment period). The area under the curve was measured for different components of the ERP including P1 and P2 (positive components) and N1 and N2 (negative components). The average area under the curve was recorded for each component at each time point and change from baseline was calculated. Individuals with FXS are thought to have excessive ERP response, so a decrease in area under each curve compared to baseline would indicate a favorable outcome.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: μV*seconds
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
μV*seconds
  P1 Component | 0.009766667 (0.001838821) | 0.010784615 (0.002861501) | 0.012972727 (0.003341777) | 0.00621 (0.001656264)
  P2 Component | 0.041122167 (0.007281467) | 0.031379615 (0.009411693) | 0.046629091 (0.009927824) | 0.0558891 (0.014525993)
  N1 Component | 0.025633667 (0.006968832) | 0.029363077 (0.006649054) | 0.035257182 (0.007841523) | 0.0354182 (0.008270948)
  N2 Component | 0.033444167 (0.009811161) | 0.038742385 (0.01309467) | 0.028213 (0.012192131) | 0.0185623 (0.009189006)

18. Secondary Outcome: Event-Related Potentials - Frontal Alpha Asymmetry at Resting State
Description: Event-Related Potentials (ERPs) enable extraction of neural responses associated with specific sensory, cognitive, or motor events from an overall EEG. EEG data was collected when the subject was in a resting state. Frontal alpha asymmetry measures differences in alpha activity level of the right and left hemisphere of the frontal lobe of the brain. ERP was performed at Baseline as well as at Week 4, Week 8, Week 12, Week 16 (end of each treatment period). Mean alpha asymmetry at resting state was recorded and change from baseline was calculated for each time point. Higher alpha asymmetry scores indicate greater alpha power in the right hemisphere, which corresponds to increased neural activity of the left hemisphere. High activity of the left frontal lobe is hypothesized to correspond with approach behaviors, and high activity of the right frontal lobe is thought to correspond to withdrawal behaviors. In this study, higher alpha asymmetry scores indicate a better outcome.
Time Frame: Baseline, Week 4 (EM Treatment), Week 8 (EM+5-HTP Treatment), Week 12 (5-HTP Treatment), Week 16 (Placebo Treatment)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Ergoloid Mesylates (EM) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | 5-hydroxytryptophan (5-HTP) | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
unitless | 0.044133817 (0.085312863) | -0.048217532 (0.094117681) | -0.133404775 (0.085879258) | 0.191055011 (0.106432066)

ADVERSE EVENTS:
Time Frame: Adverse events, which include abnormal and clinically significant clinical laboratory test variables, will be monitored and documented from the time Informed Consent until study participation is complete, 1 week after the final study visit (~21 weeks total).
Description: Participants who experience AEs will be monitored with relevant clinical assessments and laboratory tests, as determined by the Investigator. Per good medical practice, all AEs must be followed to satisfactory resolution or stabilization of the event(s), or, if a chronic condition, until fully characterized. Participants who have non-serious AEs that are ongoing at study completion or study withdrawal must be followed until resolution of the AEs or for 30 days after the last dose of study drug.
Groups:
- Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP): Ergoloid mesylates (EM) 1 mg three times daily and 5-hydroxytryptophan (5-HTP) 100 mg three times daily for 4 weeks
  5-Hydroxytryptophan / Vitamin B6: 5-hydroxytryptophan, also known as 5-HTP has a nutraceutical status and has never been approved as a drug for any indication, but as a dietary supplement has been used extensively for several disorders for many years such as in the therapy of depression, fibromyalgia, obesity, insomnia and chronic headache
  Ergoloid Mesylate: Ergoloid Mesylates, trade name Hydergine, is a mixture of the methanesulfonate salts of three dihydrogenated ergot alkaloids, dihydroergocristine, dihydroergocornine, and alpha- and beta-dihydroergocryptine. Ergot alkaloids are dopamine agonists which activate dopamine receptors (in the basal ganglia and other parts of the brain involved in motor function) and a prolactin inhibitor. Ergot is a strong vasoconstrictor and thus helps to reduce bleeding by narrowing of the blood vessels.
- Placebo: 2 placebo capsules three times daily for 4 weeks
  Placebo: Placebo capsules
- Ergoloid Mesylates (EM) and Placebo: Ergoloid mesylates (EM) 1 mg three times daily and 1 placebo capsule three times daily for 4 weeks.
  Ergoloid Mesylate: Ergoloid Mesylates, trade name Hydergine, is a mixture of the methanesulfonate salts of three dihydrogenated ergot alkaloids, dihydroergocristine, dihydroergocornine, and alpha- and beta-dihydroergocryptine. Ergot alkaloids are dopamine agonists which activate dopamine receptors (in the basal ganglia and other parts of the brain involved in motor function) and a prolactin inhibitor. Ergot is a strong vasoconstrictor and thus helps to reduce bleeding by narrowing of the blood vessels.
  Placebo: Placebo capsules
- 5-hydroxytryptophan (5-HTP) and Placebo: 5-hydroxytryptophan (5-HTP) 100 mg three times daily and 1 placebo capsule three times daily for 4 weeks.
  5-Hydroxytryptophan / Vitamin B6: 5-hydroxytryptophan, also known as 5-HTP has a nutraceutical status and has never been approved as a drug for any indication, but as a dietary supplement has been used extensively for several disorders for many years such as in the therapy of depression, fibromyalgia, obesity, insomnia and chronic headache
  Placebo: Placebo capsules
Arm/Group | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) | Placebo | Ergoloid Mesylates (EM) and Placebo | 5-hydroxytryptophan (5-HTP) and Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 3/15 | 2/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergoloid Mesylates (EM) and 5-hydroxytryptophan (5-HTP) (N=15) | Placebo (N=15) | Ergoloid Mesylates (EM) and Placebo (N=15) | 5-hydroxytryptophan (5-HTP) and Placebo (N=15)
Increased Irritability (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05030129/Prot_SAP_000.pdf